CLINICAL TRIAL: NCT06022263
Title: A Prospective, Randomised, Double-blinded, Placebo-controlled Study Investigating the Safety and Tolerability of STA363 in Patients With Radiculopathy Caused by Lumbar Disc Herniation
Brief Title: STA363 in the Treatment of Lumbar Disc Herniation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stayble Therapeutics (Industry)
Collaborators: Cromsource (Industry); Antaros Medical (Industry); VIEDOC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STA-LDH01
Record Dates: First submitted 2023-08-21; First posted 2023-09-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar radiculopathy
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy | interventions — Lactic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1.5 mL of Omnipaque mixed with water for injection
  Interventions: Drug: Placebo
- STA363 (Experimental): 1.5 mL of STA363 (lactic acid, 120 mg/mL) mixed with Omnipaque
  Interventions: Drug: Lactic Acid

INTERVENTIONS:
Drug: Lactic Acid — 180 mg of STA363 will be slowly injected into a symptom-generating herniated lumbar disc
  Other Names: STA363
  Arms: STA363
Drug: Placebo — 1.5 mL of Omnipaque in water for injection will be slowly injected into a symptom-generating herniated lumbar disc
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to establish safety and tolerability of STA363 injected into a herniated intervertebral disc in patients with sciatica due to disc herniation. The main questions the trial aims to answer are:

1. Is the treatment safe and tolerable?
2. Does the volume of the disc and the herniation decrease?
3. Is sciatica reduced? Participants will be given an injection into the herniated disc of either placebo or STA363 (one dose).

Researchers will compare safety, tolerability, effects on disc and herniation volume and on symptoms between the group of patients injected with placebo and the group injected with STA363.

DETAILED DESCRIPTION:
The study will include 24 patients, recruited at 4 different sites, suffering from radiculopathy due to lumbar disc herniation (LDH). Patients will be screened for symptoms, disease history and magnetic resonance imaging (MRI) evidence of LDH. Baseline data (e.g. pain recording and MRI data) will be collected, and 1/3 of the patients will then be randomized to intradiscal injection with placebo (Omnipaque with water for injection, 1.5 mL) and 2/3 of the patients will be randomized to STA363 (lactic acid, 120 mg/mL with Omnipaque, 1.5 mL). The injections will be done using fluoroscopic guidance, and the patients will be treated with intravenous antibiotics and sedatives. The first follow-up will be done by phone 1 week after the treatment, while the other follow-ups will be physical visits at month 1, 3 and 6 at the site. In conjunction with the visits, the patient will record daily pain intensity (Numerical Rating Scale) for 7 days using an eDiary, and MRI will be performed. The primary completion time is 6 months with the primary objectives safety and tolerability. Important secondary objectives will be changes of disc volume and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedures
2. Patient has a single subligamentous posteriolateral lumbar disc herniation (protrusion or extrusion) of any lumbar disc below L1/L2 diagnosed by clinical symptoms and/or physical findings and confirmed by MRI
3. Patient has symptoms and/or physical findings consistent with a unilateral radiculopathy affecting one nerve root (L2-L5)
4. Patient has leg pain of the dermatome consistent with the nerve root affected by the herniation
5. The herniated disc is 3 or lower on the Pfirrmann scale (grade 1-5)
6. Patient has experienced symptoms of a herniated disc for at least 6 weeks prior to randomisation without sufficient relief with pain medications and other conservative therapies
7. Ability to understand the written and verbal information about the study
8. Male and female patients 18 years or older but 50 years or younger
9. Women of childbearing potential eligible if using effective contraceptives
10. Patient has a body mass index (BMI) of ≥18 to ≤35 kg/m2
11. Patients who meet all the following NRS selection criteria for radicular leg pain:

    1. Presence of at least 5 pain NRS assessments (entries) for 7 consecutive days
    2. NRS daily pain scores between 3-9
    3. Not more than 2 NRS scores of "3"

Exclusion criteria:

1. Treatment with any investigational product within 3 months prior to the screening visit
2. Patient has a sequestered lumbar disc herniation or transligamentous/ herniation confirmed by MRI
3. Patient has a bulging disc
4. Patient has experienced symptoms of lumbar disc herniation for more than 6 months
5. Patient has 2 or more symptomatic lumbar disc herniations (presence of non-symptomatic herniations in addition to the symptomatic herniation is allowed)
6. Patient has cauda equina syndrome
7. Previous intradiscal therapeutic intervention of the index disc or has had any lumbar spine surgery
8. Presence of lumbar spine disease and/or clinically significant deformity other than a lumbar disc herniation which, in the opinion of the investigator, will affect evaluation of safety and/or efficacy
9. Untreated, ongoing active infection and/or discitis
10. Current infection or prior history of spinal infection (e.g., discitis, septic arthritis, epidural abscess) or an active systemic infection.
11. Evidence of prior lumbar vertebral body fracture or trauma.
12. Spondylolisthesis or retrolisthesis grade 2 and above or spondylolysis at the index or adjacent level(s).
13. Lumbar spondylitis or other undifferentiated spondyloarthropathy affecting the index disc.
14. Patients previously included in the study.
15. Patients suffering from psychosomatic pain in the opinion of the Investigator.
16. Patients requiring continuous treatment with warfarin or other anticoagulant therapy.
17. Known alcohol and/or drug abuse.
18. Pregnant or lactating females, or intention to become pregnant within the study period.
19. Known allergy or intolerance to the contrast agent Omnipaque®.
20. Known opioid allergy or intolerance.
21. Any other condition that, in the opinion of the Investigator, precludes the patient from taking part in this study.
22. Any specific contraindication for MRI such as claustrophobia, intracranial clips or pacemakers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Baseline and 1 week and 1,3 and 6 months after intervention for all outcomes except changes in IVD morphology (time frame 1, 3 and 6 months after intervention)
  Safety and tolerability will be measured using the following outcomes:
  * Incidence and nature of adverse events (AEs)
  * Changes in
    * physical examination findings
    * blood pressure and heart rate
    * 12-lead electrocardiogram
    * Hematology and clinical chemistry
    * Pain intensity at the injection site during and 15 minutes after injection (numerical rating scale; NRS). NRS is reported on a 0-10 scale where 0 represents "No pain" and 10 "Worst imaginable pain"
    * Other aspects of intervertebral disc morphology (IVD) morphology from baseline (e.g., Modic changes)

SECONDARY OUTCOMES:
Disc volume | Baseline and 1,3 and 6 months after intervention
  Volume will be measured by MRI
Disc height | Baseline and 1,3 and 6 months after intervention
  Height will be measured by MRI
Radicular leg pain | Baseline and 1 week and 1,3 and 6 months after intervention
  Leg pain will be reported by the patients using an NRS. (minimum value: 0; maximum value: 10) for 7 consecutive days. Lower scores means a better outcome.
Patient Global Impression of Change (PGIC) | Baseline and 1 week and 1,3 and 6 months after intervention
  PGIC will be reported by the patients using an electronic device
Disc intensity | Baseline and 1,3 and 6 months after intervention
  The intensity of the disc will be measured using T2-weighted MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jarkko Kalliomäki, MD, PhD, Study Director — Stayble Therapeutics AB
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 4, Klinika Ortopedii i Rehabilitacji, Lublin, Lublin Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No